CLINICAL TRIAL: NCT03039049
Title: GnRH Agonist Trigger and Modified Luteal Phase Support, Adding a Mid-luteal Bolus of GnRHa: a Randomised Controlled Trial.
Brief Title: GNRH Agonist Trigger and Modified Luteal Phase Adding a Bolus of GnRHa at the Time of Implantation: a RCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Ibn Rochd (Other)
Responsible Party: Principal Investigator, benmachiche abdelhamid, Dr benmachiche abdelhamid, private infertility centre, Ibn rochd, constantine, Algeria, Centre Hospitalier Universitaire Ibn Rochd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02053779
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Infertility
Keywords: GnRH agonist trigger; IVF; Luteal phase support; Mid-luteal GnRH agonist
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GnRH agonist (Experimental): Drug: Triptorelin 0.1mg Triptorelin 0.1 mg administered subcutaneously 6 days after ovum pick-up (OPU) in IVF/ICSI cycles triggered by triptorelin 0.2 mg.
  Other Names:
  • Decapeptyl 0.1 mg
  Interventions: Drug: Triptorelin 0.1 mg
- Control (No Intervention): No intervention

INTERVENTIONS:
Drug: Triptorelin 0.1 mg — a single dose of Triptorelin 0.1 mg subcutaneously administered 6 days after oocyte retrieval.
  Other Names: Decapeptyl 0.1 mg
  Arms: GnRH agonist

SUMMARY:
Purpose:The aim of this project is to prospectively determine whether a single dose of GnRH-agonist administered at the time of implantation increases or not the reproductive outcome in patients undergoing in vitro fertilization ( IVF)/ intracytoplasmatic sperm injection(ICSI) triggered by a GnRH-agonist followed by a small bolus of human chorionic gonadotropin (hCG 1500 IU) the day of oocyte retrieval.

DETAILED DESCRIPTION:
It has been reported in previous publications that the ovarian hyperstimulation syndrome (OHSS) was eliminated when GnRH agonist was used to trigger ovulation and the delivery rate has improved after modified luteal support especially when a small bolus of hCG is used on the day of oocyte retrieval. (OMEGA/HCG 1500 IU).

However, a risk difference of 7% in delivery rates is still in favor of HCG trigger. Thus, further modifications in the luteal phase supplementation are required in order to optimise the reproductive outcome after GnRH-agonist triggering.

Recently, many papers showed, that independently of the GnRH analogue used to prevent the premature LH surge, the addition of GnRH-agonist during the luteal phase seems to be beneficial in terms of pregnancy. Nevertheless, their use in practice is not yet admitted because of controversial results in terms of efficacy and safety particularly on the conceptus.

ELIGIBILITY:
Inclusion Criteria:

Female age < 40 years No uterine (fibroids, mullerian malformations), ovarian ( endometrioma) or adnexa (hydrosalpinx) abnormalities• Baseline FSH and LH < 12 IU/l.Patients with at least one embryo at transfer time

Exclusion Criteria:

* Very high risk of OHSS (> 30 follicles > 12 mm the day of ovulation triggering). • Reduced ovarian reserve

  * Fertilization failure
  * Severe endocrinopathy
  * Azoospermia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 328 (Actual)
Dates: Start 2014-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
implantation rate | Time Frame: 5 weeks after IVF/ICSI
  number of gestational sacs per number of embryos transferred

SECONDARY OUTCOMES:
positive pregnancy test | Time Frame: 2 weeks after IVF/ICSI
  confirmed by beta-hCG 14 days post embryo transfer
Ongoing pregnancy | Time Frame: 12 weeks after IVF/ICSI
  presence of foetal heart beat at 12 weeks of gestation
Delivery rate | Time Frame: 26 weeks after IVF/ICSI
  birth of baby beyond 26 weeks of gestation
Early pregnancy loss | Time Frame: miscarriage before 5 weeks of gestation
  loss of embryo before 5 weeks of gestation, chemical pregnancy and extra-uterine pregnancy

OTHER OUTCOMES:
ovarian hyperstimulation syndrome OHSS | Time Frame: from date of triggering until 2 weeks after pregnancy test]
  early and late onset Ovarian hyper stimulation syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Abdelhamid Benmachiche, M.D, Principal Investigator — Ibn roch infertility centre, cité boussouf, Constantine Algeria
Locations (2):
- Algeria (2):
  - Ibnrochd Clinic, Constantine
  - Ibnrochd IVF center, Constantine

IPD SHARING:
Plan to Share IPD: No